CLINICAL TRIAL: NCT07126925
Title: Effectiveness of an Improved Fall Risk Assessment Form Combined With Obstacle Physical Activity Testing in Preventing Falls in Elderly Hospitalized Patients
Brief Title: A Trial of an Improved Fall Risk Assessment and Activity Test to Prevent Falls in Elderly Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yang Lu, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022S0477
Record Dates: First submitted 2025-08-09; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Falls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Personalized Fall Prevention Group (Experimental): Patients in this group received universal fall precautions plus a comprehensive assessment using the "Improved Risk Assessment Form for Inpatient Falls" and the "Obstacle Physical Activity Ability Test." Based on the assessment results, a personalized fall prevention plan was developed and implemented by the nursing and physical therapy team.
  Interventions: Behavioral: Personalized Fall Prevention Program
- Active Comparator: Standard Care Group (Active Comparator): Patients in this group received the hospital's standard of care for fall prevention. This included universal fall precautions and a standard risk assessment using the hospital's existing protocol based on static factors. Interventions were standard and not explicitly tailored to individual functional deficits.
  Interventions: Behavioral: Standard Fall Prevention Care

INTERVENTIONS:
Behavioral: Personalized Fall Prevention Program — An intervention package featuring a comprehensive, multidimensional risk assessment using an improved form and a dynamic functional test (Obstacle Physical Activity Ability Test). The assessment guided the development of a personalized prevention plan, including targeted exercises, environmental adjustments, and enhanced patient/family education.
  Arms: Experimental: Personalized Fall Prevention Group
Behavioral: Standard Fall Prevention Care — Standard hospital care for fall prevention, including universal precautions (e.g., clutter-free environment, non-slip footwear) and risk assessment using a standard hospital checklist.
  Arms: Active Comparator: Standard Care Group

SUMMARY:
This randomized controlled trial was conducted to evaluate if a personalized fall prevention strategy could reduce fall incidence in elderly hospitalized patients. A total of 320 patients were randomized into two groups. The experimental group received interventions guided by an improved fall risk assessment form and an obstacle physical activity test. The control group received standard hospital care. The primary outcome was the incidence of falls. Secondary outcomes included injury severity, nursing satisfaction, patient compliance, and quality of life.

DETAILED DESCRIPTION:
Falls are a common and serious adverse event among elderly hospitalized patients. While standard risk assessment tools exist, they often fail to capture dynamic risk factors related to patient mobility and environmental interaction. This study aimed to determine if a comprehensive assessment approach could improve fall prevention outcomes. This was a single-center, randomized controlled trial. A total of 320 inpatients aged 65 and older were randomly assigned to either an experimental group or a control group. The experimental group was assessed using an "Improved Risk Assessment Form for Inpatient Falls" and a novel "Obstacle Physical Activity Ability Test." The results guided a personalized fall prevention plan, including targeted exercises and environmental modifications. The control group received the hospital's standard fall prevention care, which included a standard risk checklist and universal precautions. The study's main objective was to compare the incidence of falls between the two groups throughout their hospital stay. Other outcomes, such as injury severity, patient satisfaction, compliance with preventive measures, and quality of life, were also assessed to evaluate the broader impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients aged 65 and above.
* Identified as being at risk of falling upon admission screening (defined as having at least one of the following: history of a fall in the last 6 months, use of a walking aid, or observed gait/balance instability).
* Able to provide informed consent or have a legal guardian provide consent.

Exclusion Criteria:

* Acutely life-threatening conditions or severe cardiorespiratory instability that would preclude any mobility testing.
* History of a severe fall-related injury (defined as a fracture or head injury requiring hospitalization) in the past 6 months that currently limits mobility assessment.
* Non-ambulatory or bed-bound patients.
* Patients with severe dementia (e.g., Mini-Mental State Examination score < 10) or diagnosed psychiatric conditions (e.g., psychosis, severe agitation) that would prevent cooperation.
* Expected hospital stay of less than 48 hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Fall Incidence | Through study completion, an average of 10 days
  The proportion of patients experiencing one or more falls. A fall was defined as an event which results in a person coming to rest inadvertently on the ground or floor or other lower level. It was recorded through the hospital's incident reporting system, patient self-report, and daily nursing checks.

SECONDARY OUTCOMES:
Severity of Fall-Related Injury | Through study completion, an average of 10 days
  Classification of injuries sustained from a fall, categorized by a physician as: no injury, minor injury (e.g., bruises, abrasions), or major injury (e.g., fracture, head injury with loss of consciousness, laceration requiring sutures).
Nursing Satisfaction | At discharge (an average of 10 days post-admission)
  Patient-reported satisfaction with nursing communication, responsiveness, and fall prevention education, measured using a 5-item institutional survey on a 10-point scale.
Patient Compliance | Through study completion, an average of 10 days (assessed weekly)
  Adherence to prescribed fall prevention precautions, assessed via a 10-item observational checklist of precautions (e.g., using call bell, bed in low position). Compliance was categorized based on the percentage of items adhered to.
Change in Physical Activity Ability | Baseline and at discharge (an average of 10 days)
  Change in physical mobility from admission to discharge, categorized by the treating physical therapist as "Improved markedly," "Improved," "No change," or "Reduced," based on clinical judgment and performance on the obstacle test.
Change in Quality of Life (QoL) | Baseline and at discharge (an average of 10 days)
  Change in QoL from admission to discharge, measured by the mean change in a 10-point global QoL rating from a structured, non-validated questionnaire covering physical, psychological, and social domains. The scale is a 10-point global Quality of Life rating questionnaire, with a range from 1 (worst possible quality of life) to 10 (best possible quality of life). A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China